CLINICAL TRIAL: NCT04324385
Title: Accuracy of Pulse Oximeters With Profound Hypoxia
Status: Completed | Type: Observational
Sponsor: Compumedics Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: SOMFIT01
Record Dates: First submitted 2020-03-23; First posted 2020-03-27 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Oximetry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To test the accuracy of a non-invasive blood oxygen saturation monitor which is placed on a subject with profound hypoxia.

DETAILED DESCRIPTION:
A radial arterial cannula was placed in either the left or right wrist of each subject for arterial blood sampling and blood pressure monitoring. Blood gas analysis to determine oxyhemoglobin saturation (SaO2)was performed using an ABL-90 multi-wavelength oximeter (Hemoximeter, Radiometer, Copenhagen, serial 1393-090R0359N0002). This instrument contains factory certified calibration standards and quality control algorithms.

Each subject had two control blood samples taken at the beginning of each experiment, while breathing room air. Hypoxia was then induced to different and stable levels of oxyhemoglobin saturation (between 70-100%) by having subjects breathe mixtures of nitrogen, room air, and carbon dioxide. Each plateau level of oxyhemoglobin saturation was maintained for at least 30 seconds or until reference pulse oximeters readings were stable. Two arterial blood samples were then obtained, approximately 30 seconds apart. Each stable plateau therefore was maintained for at least 60 seconds with SpO2 fluctuating by less than 2-3%. The plateaus were nominally at 100%, room air saturation, 93%, 90%, 87%, 85%, 82%, 80%, 77%, 75% and 70%. A total of 270 samples were obtained at the saturation plateaus across this span. Data were provided for analysis. At least 200 data points were collected for each type of oximeter and probe combination studied.

Pulse oximeter data is taken as 5 second averages corresponding to the point of arterial blood analysis. Individual data points may be missed or excluded for dropped signals or failure of the oximeter signal to achieve an appropriate plateau. Data is plotted as Hemoximeter data (SaO2) vs. pulse oximeter bias (SpO2 - SaO2). A different marker is used for each study subject. Linear regression is shown for all subjects combined, and the equation with R2 is shown on the plot. Mean bias is displayed as a solid horizontal line, and the upper and lower limits of agreement (mean bias ± 1.96•SD*) are shown by dashed horizontal lines. For the "pooled" plots, different markers are used for each pulse oximeter. Tables of mean, standard deviation, standard error, minimum, maximum, 95% confidence interval, count and root mean square are provided for each oximeter's bias, and all oximeters combined in the following ranges of SaO2 (Hemoximeter): 60 - 80%, 80 - 100%, 60 - 100%, 70 - 100%, 50 - 60%, 60 - 70%, 70 - 80%, 80 -90%, and 90 - 100%.

ELIGIBILITY:
Inclusion Criteria:

* Normal hemoglobin levels (Hemoglobin ≤ 10gm•dl-1)
* Healthy
* Non-smoking individuals
* 21-49

Exclusion Criteria:

* Unhealthy

Ages: 21 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All of the subjects enrolled in the study had normal hemoglobin levels (Hemoglobin ≤ 10gm•dl-1) and all were healthy non-smoking individuals of age 21-49.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2019-04-09 (Actual); Primary Completion 2019-04-10 (Actual); Study Completion 2019-04-10 (Actual)

PRIMARY OUTCOMES:
Testing the accuracy of a new pulse oximeter device | Approx. 60 mins per subject
  The primary outcome measure was to find the agreement between methods of measurement with multiple observations per individual. Spo2 readings from the test device were compared with a factory certified and calibrated oxyhemoglobin saturation monitor (i.e. ABL-90 multi-wavelength oxiemter) and two other standard oximeter devices using root mean squared error as the measure of accuracy.

CONTACTS AND LOCATIONS:
Locations (1):
- Hypoxia Lab, San Francisco, California, United States